CLINICAL TRIAL: NCT03764878
Title: MARS: Magnetic Resonance Study: A Novel Assessment of Placental Function
Status: Completed | Type: Observational
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Beth Plunkett, Clinical associate professor, Endeavor Health
Other Study IDs: EH18-300
Record Dates: First submitted 2018-11-29; First posted 2018-12-05 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Placenta Diseases
MeSH Terms: conditions — Placenta Diseases | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Maternal and fetal cord plasma. Placental extracts. Formalin-fixed placental specimens.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal weight: BMI 18.5-24.9 kg/m^2 low risk pregnancy
  Interventions: Diagnostic Test: functional MRI
- Pregestational diabetes mellitus: Type 1 or Type 2 diabetes mellitus diagnosed prior to the pregnancy or in the first trimester
  Interventions: Diagnostic Test: functional MRI
- Obese: Pre-pregnancy BMI ≥ 30.0 kg/m^2
  Interventions: Diagnostic Test: functional MRI

INTERVENTIONS:
Diagnostic Test: functional MRI — Participants will undergo a functional MRI using multiple imaging modalities.

SUMMARY:
The objective of this study is to evaluate functional MRI as a tool to study placental transfer of oxygen and nutrients during the third trimester of pregnancy in obese women, women with pregestational diabetes and healthy low risk women without these conditions (controls). The investigators hypothesize that altered placental function, including diminished placental oxygenation and enhanced placental transport of lipids and metabolites will be seen in obese and pregestational diabetics as compared to controls.

DETAILED DESCRIPTION:
In this study, we propose to utilize two novel and innovative non-invasive tools to measure placental oxygenation and lipid and nutrient transport in vivo in women who are obese (OB), have pregestational diabetes (DM) or have neither (controls). To evaluate differences in placental oxygenation, we propose to use Blood Oxygen Level Depending (BOLD) imaging, a method of functional magnetic resonance imaging, to measure tissue oxygenation in the placenta during the third trimester of pregnancy. To evaluate placental lipid and nutrient content, we propose to utilize Magnetic Resonance Spectroscopy (MRS), a novel and powerful tool to compare lipid and nutrient transport across the placenta among OB, DM and controls.

To confirm in vivo BOLD and MRS findings, we will extensively evaluate the placental lipid content and lipid transport capability. Fatty acid transport protein-4 (FATP-4), one of 6 FATP proteins, is important for placental lipid accumulation, especially LC-PUFA21-24. Docosahexaenoic acid (DHA) is a crucial LC-PUFA for neurogenesis in early development18. Major facilitator super family domain containing MFSD2a is a lysophospholipid transporter required for DHA uptake in the brain and has been linked to placental DHA transfer. Lipid content of the placenta can be assessed by visualizing lipid droplets via perilipin 2, the most abundant structural protein on the surface of lipid droplets of adipocytes.

We hypothesize that altered placental function including diminished placental oxygenation and abnormal placental transport of lipids and other metabolites will be seen in OB and DM women as compared to controls. We further hypothesize that ex vivo placental pathologic, histologic and immunohistochemistry characteristics will be associated with in vivo findings. Our findings from this pilot study have the potential to serve as the basis of a larger study to further evaluate the potential impact of BOLD and MRS technology on our understanding of placental lipid and oxygen transport among women with obesity and pregestational diabetes as compared to women without these conditions.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* planned cesarean section

Exclusion Criteria:

* non-English speaking
* fetal anomalies
* gestational diabetes mellitus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women at 30-34 weeks gestation who are scheduled for a cesarean delivery. For this pilot project, 10 obese (OB) women, 10 women with pregestational diabetes (PGD) and 10 women without OB or PGD will be recruited. OB is defined as prepregnancy or first trimester BMI greater than or equal to 30 kg/ m2. PGD will be defined as Type 1 or Type 2 diabetes diagnosed prior to the pregnancy or in the first trimester.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Change in BOLD response level in the placenta | 1 day
  As measured by the change in MRI from baseline (room air) compared to hyperoxygenation (O2 facemask) in the central area of the placenta

SECONDARY OUTCOMES:
Placenta ratio of oxygenated hemoglobin to deoxygenated hemoglobin | 1 day
  As measured on MRI during third trimester in the central area of the placenta
Placenta ratio of choline to lipid | 1 day
  As measured on MRI during third trimester in the central area of the placenta

CONTACTS AND LOCATIONS:
Overall Officials: Beth Plunkett, MD, MPH, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided